CLINICAL TRIAL: NCT00328861
Title: Phase II Study in Metastatic Melanoma or Kidney Cancer Using Autologous Natural Killer Cells Plus Aldesleukin (IL-2) Following a Lymphodepleting Chemotherapy
Brief Title: Natural Killer Cells Plus IL-2 Following Chemotherapy to Treat Advanced Melanoma or Kidney Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Steven A. Rosenberg, M.D./National Cancer Institute, National Institutes of Health
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 060169; 06-C-0169; NCT00354055 (obsolete NCT alias)
Record Dates: First submitted 2006-05-20; First posted 2006-05-22 (Estimated); Results first posted 2012-11-05 (Estimated); Last update posted 2012-11-05 (Estimated); Status verified 2012-10

CONDITIONS: Metastatic Melanoma; Metastatic Kidney Cancer
Keywords: Adoptive Cell Therapy; Cutaneous Melanoma; Clinical Response; Rate of Repopulation; Toxicity Profile; Metastatic Melanoma; Metastatic Kidney Cancer
MeSH Terms: conditions — Melanoma; Kidney Neoplasms | interventions — Lymphocyte Count; Interleukin-2; aldesleukin; Cyclophosphamide; fludarabine; fludarabine phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- NK Cells + IL-2: Melanoma (Experimental): Melanoma (skin cancer). Cyclophosphamide 60 mg/kg/day intravenous on days -8 and -7. Fludarabine 25 mg/m^2 day intravenous on days -6 through -2. IL-2 720,000 IU/kg/intravenous every 8 hours for up to 5 days. Thirty minutes infusion of natural killer (NK) cells 2 days after last dose of chemotherapy.
  Interventions: Drug: Natural Killer (NK) Lymphocytes; Biological: IL-2; Drug: Cyclophosphamide; Drug: Fludarabine
- NK Cells + IL-2: Renal Cell (Experimental): Renal cell (kidney cancer). Cyclophosphamide 60 mg/kg/day intravenous on days -8 and -7. Fludarabine 25 mg/m^2 day intravenous on days -6 through -2. IL-2 720,000 IU/kg/intravenous every 8 hours for up to 5 days. Thirty minutes infusion of natural killer (NK) cells 2 days after last dose of chemotherapy.
  Interventions: Drug: Natural Killer (NK) Lymphocytes; Biological: IL-2; Drug: Cyclophosphamide; Drug: Fludarabine

INTERVENTIONS:
Drug: Natural Killer (NK) Lymphocytes — Thirty minutes infusion of natural killer (NK) cells 2 days after last dose of chemotherapy.
  Other Names: NK cells
Biological: IL-2 — IL-2 720,000 IU/kg/intravenous every 8 hours for up to 5 days.
  Other Names: aldesleukin
Drug: Cyclophosphamide — Cyclophosphamide 60 mg/kg/day intravenous on days -8 and -7.
  Other Names: Cytoxan
Drug: Fludarabine — Fludarabine 25 mg/m^2 day intravenous on days -6 through -2.
  Other Names: Fludara

SUMMARY:
Background:

* Natural killer (NK) cells are large lymphocytes (a type of white blood cell) that are important in the immune response to cancer.
* IL-2 (Aldesleukin) is a substance the body makes that controls the growth and function of many types of cells. The Food and Drug Administration has approved IL-3 for treating metastatic melanoma and kidney cancer. (Metastatic disease is cancer that has spread beyond the primary site.)

Objectives: To determine the safety and effectiveness of treating metastatic melanoma and kidney cancer with laboratory-treated NK cells and IL-2.

Eligibility: Patients 18 years of age or older with metastatic melanoma or kidney cancer who have previously been treated with high-dose IL-2.

Design:

* Leukapheresis. Patients under leukapheresis to obtain NK cells for the treatment regimen. Blood is collected through a needle in an arm vein and directed through a cell separator machine where white blood cells are extracted. The rest of the blood is returned to the patient through a needle in the other arm. NK cells are removed from the white blood cells and treated for re-infusion into the patient.
* Chemotherapy. Starting 8 days before infusion of the treated NK cells, patients receive intravenous (IV, through a vein) infusions of cyclophosphamide and fludarabine to suppress the immune system.
* NK cell infusion. Patients receive a 30-minute IV infusion of NK cells 2 days after the last dose of chemotherapy.
* IL-2 therapy. Within 24 hours of the NK cell infusion, patients receive high-dose IL-2 as a 15-minute IV infusion every 8 hours for up to 5 days. A second cycle of IL-2 is given about 14 days after the first.
* Blood tests and biopsy. Patients have frequent blood tests during the treatment period and may be asked to undergo a biopsy (surgical removal of a small piece of tumor or lymph node) at the end of treatment to look at the effects of the treatment on the tumor immune cells.
* Follow-up evaluation. Patients are evaluated 4-6 weeks after completing treatment. They have a physical examination, scans of tumor sites, blood tests and blood sampling (or leukapheresis) to examine the response to treatment. Patients who improve with treatment return for evaluations every month. Those whose tumor grows again after originally shrinking may receive one additional treatment course.

DETAILED DESCRIPTION:
Background:

* Natural killer (NK) cells are large granular lymphocytes that are critical effector cells in the early innate immune response to pathogens and cancer.
* Previous and current clinical investigations have clearly demonstrated that T lymphocytes can mediate the regression of metastatic melanoma. However, not all patients with cancer are eligible for this type of immunotherapy either because resectable tumor is not available, the TIL do not expand sufficiently, or the tumor infiltrating lymphocytes (TIL) that do proliferate do not exhibit sufficient tumor specific reactivity.
* We have recently developed techniques for the in vitro isolation and expansion of anti-tumor NK cells to levels suitable for the treatment of cancer patients and are proposing in this protocol to evaluate therapy using these NK cells.
* In Surgery Branch pre-clinical experiments, we evaluated lysis of fresh melanoma cell digests, melanoma cell lines, renal cell carcinoma (RCC) lines, and normal peripheral blood mononuclear cells (PBMCs) by NK cells from several patients and demonstrated that NK cells could lyse some fresh melanoma digests, as well as melanoma cell lines and renal cell cancer (RCC) lines, while sparing normal allogeneic and autologous PBMCs.

Objectives:

* Determine the ability of the administration of autologous natural killer (NK) cells plus aldesleukin (IL-2) following a non-myeloablative lymphodepleting preparative regimen to mediate tumor regression in patients with metastatic melanoma or kidney cancer.
* Determine the rate of repopulation of the natural killer cells in treated patients.
* Determine the toxicity of this treatment regimen.

Eligibility:

* Patients, 18 years of age or older with metastatic melanoma or metastatic kidney cancer who have previously received high dose IL-2, with an Eastern Cooperative Oncology Group (ECOG) of 0 or 1.
* Patients may not have any active systemic infections, coagulations disorders, major medical illnesses of the cardiovascular, respiratory or immune systems or any form of autoimmune disease or immunodeficiency.

Patients must be eligible to receive high-dose IL-2.

Design:

* Patients will undergo apheresis on 03-C-0277 (Cell Harvest and Preparation for Surgery Branch Adoptive Cell Therapy Protocols) to obtain cells for generation of autologous natural killer cells.
* All patients will receive a non-myeloablative lymphocyte depleting preparative regimen of cyclophosphamide (60 mg/kg/day IV) on days -8 and -7 and fludarabine (25 mg/m^2/day IV) on days -6 through -2.
* On day 0 patients will receive the infusion of autologous natural killer lymphocytes and then begin the first cycle of high-dose IL-2 (720,000 IU/kg IV every 8 hours for up to 15 doses). A second cycle of IL-2 will be administered approximately 14 days later.
* Clinical and Immunologic response will be evaluated about 4 to 6 weeks

after the second cycle of IL-2.

-Using a small optimal Phase II design, two cohorts of patients, initially 16 in each cohort, will be enrolled, and if at least one of the first 16 patients has a clinical response (partial response (PR) or complete response (CR)), accrual will continue to 29 patients, targeting a 15% goal for objective response.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Patients must have previously received high dose IL-2 (aldesleukin) and have been either non-responders (progressive disease) or have recurred.
  2. Patients who are greater than or equal to 18 years of age, must have measurable metastatic melanoma or metastatic kidney cancer and no tumor reactive T cells available for cell transfer therapy.
  3. Pathology for metastatic melanoma or metastatic kidney cancer to be confirmed by the National Cancer Institute (NCI) Laboratory of Pathology.
  4. Patients of both genders must be willing to practice birth control for four months after receiving the preparative regimen.
  5. Clinical performance status of Eastern Cooperative Oncology Group (ECOG) 0, 1.
  6. Absolute neutrophil count greater than 1000/mm^3.
  7. Platelet count greater than 100,000/mm^3.
  8. Hemoglobin greater than 8.0 g/dl.
  9. Serum alanine aminotransferase (ALT)/aspartate aminotransferase (AST) less than three times the upper limit of normal.
  10. Serum creatinine less than or equal to 1.6 mg/dl.
  11. Total bilirubin less than or equal to 2.0 mg/dl, except in patients with Gilbert's Syndrome who must have a total bilirubin less than 3.0 mg/dl.
  12. Must be willing to sign a durable power of attorney.

EXCLUSION CRITERIA:

1. Less than four weeks has elapsed since any prior systemic therapy at the time the patient receives the preparative regimen, or less than six weeks since prior nitrosurea therapy.
2. Women of child-bearing potential who are pregnant or breastfeeding because of the potentially dangerous effects of the preparative chemotherapy on the fetus or infant.
3. Life expectancy of less than three months.
4. Systemic steroid therapy required.
5. Any active systemic infections, coagulation disorders or other major medical illnesses of the cardiovascular, respiratory or immune system, as evidenced by a positive stress thallium or comparable test, myocardial infarction, cardiac arrhythmias, obstructive or restrictive pulmonary disease.
6. Any form of autoimmune disease (such as autoimmune colitis or Crohn's Disease).
7. Seropositive for human immunodeficiency virus (HIV) antibody. (The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who are HIV seropositive can have decreased immune competence and thus be less responsive to the experimental treatment and more susceptible to its toxicities.)
8. Seropositive for hepatitis B or C antigen.
9. Seronegative for Epstein-Barr virus (EBV).
10. Patients who are not eligible to receive high-dose Aldesleukin as evaluated by the following:

    1. Patients who are 50 years old or greater who do not have a normal stress cardiac test (stress thallium, stress multi-gated acquisition scan (MUGA), dobutamine echocardiogram, or other stress test) will be excluded.
    2. Patients who have history of electrocardiogram (EKG) abnormalities, symptoms of cardiac ischemia or arrhythmias who do not have a normal stress cardiac test (stress thallium, stress MUGA, dobutamine echocardiogram, or other stress test) will be excluded.
    3. Patients with a prolonged history of cigarette smoking or symptoms of respiratory dysfunction who do not have a normal pulmonary function test as evidenced by a forced expiratory volume 1 (FEV1) less than 60% predicted will be excluded.
    4. Patients who experienced toxicities during prior IL-2 administration that would preclude redosing with IL-2, i.e. myocardial infarction, mental status changes requiring intubation, bowel perforation or renal failure requiring dialysis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2006-05; Primary Completion 2007-07 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute (NCI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Berendt MJ, North RJ. T-cell-mediated suppression of anti-tumor immunity. An explanation for progressive growth of an immunogenic tumor. J Exp Med. 1980 Jan 1;151(1):69-80. doi: 10.1084/jem.151.1.69. PMID 6444236
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/detail/A_2006-C-0169.html

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | NK Cells + IL-2: Melanoma | NK Cells + IL-2: Renal Cell
Started | 7 | 1
Completed | 7 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | NK Cells + IL-2: Melanoma | NK Cells + IL-2: Renal Cell | Total
Number analyzed (Participants) | 7 | 1 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 1 | 8
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 37.3 (11.0) | 51.0 (0) | 39.0 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 0 | 4
  Male | 3 | 1 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 7 | 1 | 8
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 7 | 1 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 1 | 8

OUTCOME MEASURES:

1. Primary Outcome: Objective Response
Description: Objective response (complete response (CR) or partial response (PR)) is measured by the Response Evaluation Criteria in Solid Tumors (RECIST) criteria. Complete response (CR) is the disappearance of all target lesions. Partial response (PR) is at least a 30% decrease in the sum of the longest diameter (LD) of target lesions taking as reference the baseline sum LD.
Time Frame: very 4-6 weeks for up to 1 year, and then every 6 months for up to 5 years.
Measure: Number; unit: Participants
Arm/Group | NK Cells + IL-2: Melanoma | NK Cells + IL-2: Renal Cell
Number analyzed (Participants) | 7 | 1
Participants
  Complete Response | 0 | 0
  Partial Response | 0 | 0

2. Secondary Outcome: Safety
Description: Here is the number of participants with adverse events. For the detailed list of adverse events see the adverse event module.
Time Frame: 11/30/2006 - 7/31/2007
Measure: Number; unit: Participants
Arm/Group | NK Cells + IL-2: Melanoma | NK Cells + IL-2: Renal Cell
Number analyzed (Participants) | 7 | 1
Participants | 7 | 1

ADVERSE EVENTS:
Arm/Group | NK Cells + IL-2: Melanoma | NK Cells + IL-2: Renal Cell
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/1
Other Adverse Events (participants affected / at risk) | 7/7 | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NK Cells + IL-2: Melanoma (N=7) | NK Cells + IL-2: Renal Cell (N=1)
Leukocyte count decreased (Blood and lymphatic system disorders) | 7 (7) | 1 (1)
Lymphocyte count decreased (Blood and lymphatic system disorders) | 7 (12) | 1 (2)
Neutrophil count decreased (Blood and lymphatic system disorders) | 7 (7) | 1 (1)
Platelet count decreased (Blood and lymphatic system disorders) | 7 (7) | 1 (1)
Hypotension (Cardiac disorders) | 1 (1) | 1 (1)
Activated partial thromboplastin time prolonged (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Fatigue (General disorders) | 6 (8) | 1 (2)
Nausea (Gastrointestinal disorders) | 6 (8) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (4) | 1 (1)
Petechiae (Blood and lymphatic system disorders) | 4 (4) | 1 (1)
Hemorrhage nasal (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Serum albumin decreased (Metabolism and nutrition disorders) | 4 (4) | 1 (1)
Serum phosphate decreased (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Confusion (Nervous system disorders) | 3 (4) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (3)
Capillary leak syndrome (Vascular disorders) | 5 (6) | 1 (1)
Hemoglobin decreased (Blood and lymphatic system disorders) | 3 (3) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Premature ventricular contractions (Cardiac disorders) | 1 (1) | 0 (0)
Fever (General disorders) | 2 (2) | 0 (0)
General symptom (General disorders) | 2 (2) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash desquamating (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Anorexia (Gastrointestinal disorders) | 1 (2) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 2 (3) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 1 (2) | 0 (0)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 2 (3) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 1 (2) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Serum calcium decreased (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Serum potassium decreased (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Serum sodium decreased (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Blood uric acid increased (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Chest pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pain in extremity (General disorders) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 4 (7) | 0 (0)
Neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 0 (0)
Bilirubin increased (Metabolism and nutrition disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No